CLINICAL TRIAL: NCT07299175
Title: Assessment of Digital Mental Integrated Intervention Technology on Language Improvement in Children of Autism: One Centre Study
Brief Title: Digital Mental Integrated Intervention Technology on Language Improvement on Autistic Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Makari masri isaac mousa, Master student in Pediatric Department, Ain Shams University
Other Study IDs: technology effect on ASD child
Record Dates: First submitted 2024-09-20; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: application called Mental Imagery Therapy for Autism (MITA) — If an application called Mental Imagery Therapy for Autism (MITA) has an effect on language improvement,sociability and cognitive awareness in a sample of children with Autism to seek to provide a tablet-based therapeutic application as a means of reducing the therapy gap and improve quality of care .

SUMMARY:
Primary aim: evaluate the effect of MITA application on language improvement in children with Autism.

Secondary aim: evaluate the effect of MITA application on sociability and cognitive awareness in children with Autism.

DETAILED DESCRIPTION:
One of the most important behavioral and developmental features that suggest autism is language delays and deviations, so that social communication and social interaction is a real challenge during management of ASD patients.

Among individuals diagnosed with autism spectrum disorder ASD, the prevalence of prefrontal synthesis (PFS) paralysis is 30 to 40% ,and may be as high as 60% among children enrolled into special ASD schools The management of ASD is mainly non-pharmacological like cognitive, behavioral, speech therapy which may help to maximize communication skills The use of technology in the delivery of much needed therapy called digital therapeutics promises to be effective for shrinking the gap between the therapy that is recommended for children with ASD and the amount they receive. There has been a promising trend towards computer-based interventions which capitalize on the often observed preference children with ASD show for flat screen information.

Mental imaginary therapy for autism MITA application hypothesized to be used in early PFS-targeting intervention can improve language ability in children with ASD .

ELIGIBILITY:
Inclusion Criteria:

1. Age: 2 year to 8 years.
2. Both sexes
3. Diagnosed with autism spectrum disorders

Exclusion Criteria:

* A history of other developmental disorders or neuropsychiatric disease.

Ages: 8 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A sample of Children with ASD who were diagnosed by Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
evaluate the effect of MITA application on language improvement in children with Autism. | baseline , after 3 months and after 6 months .
  evaluation through :Autism Treatment Evaluation Checklist and Mental Synthesis Evaluation Checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd EL-Adl El-Sawy, Professor of Pediatrics, Study Chair — Professor of Pediatrics ain shams university; Ola Ali Khalifa, professor, Study Director — professor of medical genitics ain shams university; Azza Mohamed Youssef, professor, Study Director — Professor of developmental and behavioral pediatrics ain shams university; Asmaa Wafeek Abdelaziz, assistant professor, Principal Investigator — assistant prfessor of pediatrics ain shams university; Sarah Farid Mohamed Fahmy, Associate Proffessor, Principal Investigator — associate Professor of clinical pharmacy ain shams university
Locations (1):
- Ain Shams University, Cairo, Egypt